CLINICAL TRIAL: NCT05260606
Title: Imaging Biomarkers for Immune Checkpoint Inhibitor Treatment in Patients With Non-small Cell Lung Cancer: Prospective Observational Study
Brief Title: Imaging Biomarkers for Immune Checkpoint Inhibitor Treatment in Patients With Non-small Cell Lung Cancer
Acronym: IBFIC
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Ho Yun Lee, Associate professor, Samsung Medical Center
Other Study IDs: SMO1220071
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Immune Checkpoint Inhibitors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Patients with NSCLC who will have FDG PET/CT before and during ICI Tx: There is no difference from the treatment schedule performed in usual clinical setting except for an additional F-18 FDG PET/CT scan. Detailed plan of ICI treatment and patient management (dose, administration date, treatment period, and follow-up) follows the standard protocol of our institution in this study.
  Interventions: Diagnostic Test: F-18 FDG PET/CT

INTERVENTIONS:
Diagnostic Test: F-18 FDG PET/CT — 1. 1st scan: pre-Tx, ICI Tx must be started within 35 days after 1st scan.
  2. 2nd scan: interim
     * Pembrolizumab or atezolizumab: after the 2nd Tx cycle to before the start of the 3rd Tx cycle
     * Nivolumab: after the 3rd Tx cycle to before the start of the 4th Tx cycle
  3. 3rd scan: optional (3rd scan can be performed when disease progression is suspected)
  4. Imaging
     * Fasting: at least 6 hours
     * Blood glucose level: < 200 mg/dL
     * F-18 FDG 0.14 mCi/kg (IV)
     * Image acquisition: 1 hr after FDG injection, CT images are acquired. After CT scan, PET images are acquired and attenuation-corrected PET images are reconstructed based on the CT image data.
     * PET/CT: Discovery MIDR or MI (GE Healthcare, Chicago, Illinois, USA)
     * First and second scans have to be performed with same scan.

SUMMARY:
1. Hypothesis : imaging biomarkers of tumor measured by F-18 fluorodeoxyglucose (FDG) positron emission tomography(PET)/computed tomography(CT) is correlated with immune checkpoint inhibitor (ICI) treatment response and patient prognosis.
2. Purpose: To evaluate the association between metabolic imaging parameters measured by F-18 FDG PET/CT and clinical outcomes in patients with non-small cell lung cancer treated with ICIs.
3. Study subject: patients with non-small cell lung cancer who will be treated with ICIs.
4. Study design: prospective observational study
5. Intervention: F-18 FDG PET/CT

DETAILED DESCRIPTION:
1. Study purposes

1. Primary purpose: To evaluate the association between metabolic imaging parameters measured by F-18 FDG PET/CT and treatment response in non-small cell lung cancer (NSCLC) patients treated with ICIs.
2. Secondary purpose: To evaluate the association between PET imaging parameters, patient prognosis, CT imaging parameters, and other biomarkers, and to compare treatment response evaluation criteria.

2. Background: development of ICIs opened a new paradigm for cancer treatment. It enables long-term survival of patients with advanced cancers, which could not be expected to be effective with conventional chemotherapy. Therapeutic response and prognosis to ICIs have unique characteristics which are different from those of conventional cytotoxic or targeted therapies. Even if the initial response rate is not high, if the treatment effect is effective, the effect is long-lasting and enabling long-term survival. With the evaluation criteria based on the change in tumor size, it is difficult to differentiate between an atypical response of ICIs and disease progression. Therefore, a new type of approach is required. F-18 FDG PET/CT is an imaging method that is currently used for many cancers. In recent studies on the response evaluation of ICIs using FDG PET/CT, FDG PET/CT has shown potential as a predictive tool of therapeutic response and prognosis. However, despite the potential, most of the related studies are retrospective design and small in scale. Additionally, it is not known which PET imaging features are suitable for predicting treatment response and prognosis. A novel image analysis method based on image informatics has been tried. After extracting image features from imaging modalities such as PET, CT, MRI, they are fused with clinical information and genetic information and analyzed through an artificial intelligence-based platform. It has been reported that a predictive model based on CT image features can predict the treatment response to ICI. However, the efficacy of imaging biomarkers for predicting ICI treatment response has not yet been proven, and further prospective studies are needed. Therefore, patients with NSCLC to be treated with ICI will receive FDG PET/CT before and during treatment in this study. In addition, PET images will be comprehensively analyzed together with other image data, biomarkers, and clinical data, and will be used as basic data for future ICI prediction models.

3. Study design: single institution, single-arm, prospective observational study

4. Study population: NSCLC patients who are scheduled to receive ICI in our institution

5. Recruitment: clinical referrals

6. Target number: 100 patients available for analysis.

7. Intervention: F-18 FDG PET/CT scan

7. Study protocol

1. Study participants will have FDG PET/CT before and during ICI Tx.
2. There is no difference from the treatment schedule performed in usual clinical setting except for an additional F-18 FDG PET/CT scan. Detailed plan of ICI treatment and patient management (dose, administration date, treatment period, and follow-up) follows the standard protocol of our institution in this study.
3. Scans: 1st scan (pre-treatment), 2nd scan (interim), 3rd scan (Optional)

8. Variables

1. Death status, date of death
2. Disease progression status, date of disease progression
3. ICI type and dose
4. First day of ICI treatment, end day of ICI treatment, ICI treatment cycle
5. Hospital visit dates
6. Neutrophil to lymphocyte ratio (NLR)
7. Immunochemical staining results [PD-L1: Combined positive score (CPS) and tumor proportion score (TPS)]
8. Other blood and biopsy results
9. FDG PET/CT imaging parameters [Standard uptake value (SUV)max, SUVpeak, metabolic tumor volume (MTV), total lesion glycolysis (TLG), spleen to liver ratio (SLR), etc]
10. CT imaging parameters
11. PET-based treatment response: positron Emission Tomography Response Criteria in Solid Tumors (PERCIST) criteria/ immune PERCIST (iPERCIST)/ Deauville score
12. CT-based treatment response: response Criteria in Solid Tumors (RECIST v1.1) criteria / immune RECIST (iRECIST) criteria / immune-modified RECIST (imRECIST)

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or over
2. pathologically proven non-small cell lung cancer: adenocarcinoma or squamous cell carcinoma
3. patients to be treated with immune checkpoint inhibitors (nivolumab or pembrolizumab or atezolizumab)
4. ECOG performance status ≤ 2
5. A person who have heard the detailed explanation of this clinical trial and are willing to voluntarily decide to participate and sign the informed consent form

Exclusion Criteria:

1. subjects without measurable lesion: They must have at least one measurable lesion with a diameter of 10 mm by spiral CT or multi-detector CT (MD CT) or 20 mm or larger by conventional CT.
2. subjects with a history of other malignant diseases within the past 5 years, except for treated basal cell carcinoma of the skin, carcinoma in situ of the cervix, cured thyroid cancer, and early gastric cancer
3. subjects with clinically significant uncontrolled seizures, central nervous system disease, or psychiatric disorders that, in the investigator's judgment, interferes with or is likely to interfere with the understanding of informed consent
4. subjects with uncontrolled diabetes
5. subjects with severe uncontrolled infection
6. subjects who underwent major surgery within 4 weeks prior to the start of the clinical trial or who have not fully recovered from the effects of major surgery
7. pregnant or lactating patients
8. subjects who have not received a pregnancy test or have a positive result during the basic test (menopause women with amenorrhea period of at least 12 months or longer are considered infertile subjects)
9. women or men of childbearing potential who are unwilling to use contraception during the clinical trial period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years old or over with non-small cell lung cancer who will be treated with immune checkpoint inhibitors
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between metabolic imaging parameters and treatment response | The primary analysis can be performed when all study subjects have elapsed more than 6 months after the start of treatment.
  * Analyze the correlation between metabolic imaging indicators (SUVmax, SULpeak, MTV, TLG, SLR of tumor lesions on 1st scan, % change of SUVmax, % change of SULpeak, % change of MTV, % change of TLG, % change of SLR between 1st and 2nd scans) and treatment response.
  * Treatment response: If the patient maintains a stable disease state or above based on the CT response evaluation criteria for more than 6 months, it is considered to have a response.
  * % change = [((Value of SCAN2 - value of SCAN1)/value of SCAN1) X 100]
  * Analysis model: point-biserial correlation analysis (Two-tailed test)

SECONDARY OUTCOMES:
Correlation between metabolic imaging parameters and patient prognosis | The primary analysis can be performed when all study subjects have elapsed more than 12 months after the start of treatment.
  - Analyze the correlation between the metabolic imaging indicators and patient's overall survival (OS) and progression free survival (PFS) using Cox proportional hazard model
Comparison of clinical outcome according to FDG PET/CT evaluation criteria (PERCIST vs. iPERCIST) | The primary analysis can be performed when all study subjects have elapsed more than 12 months after the start of treatment.
  - Compare clinical outcome according to the FDG PET/CT evaluation criteria (PERCIST vs. iPERCIST) using Pearson chi-square test
Correlation between metabolic imaging parameters and CT imaging parameters obtained from contrast-enhanced CT | Analysis can be performed at the time when all target subjects underwent pre-treatment and interim F-18 FDG PET/CT scans.
  - Analyze the correlation between PET parameters and contrast CT parameters using Pearson or Spearman correlation analysis
Comparison of FDG PET/CT evaluation criteria with CT evaluation criteria (iRECIST and imRECIST) | Analysis can be performed at the time when all target subjects underwent pre-treatment and interim F-18 FDG PET/CT scans.
  - Compare FDG PET/CT evaluation criteria and CT evaluation criteria using Pearson chi-square test
Correlation between imaging markers and non-imaging biomarkers | Analysis can be performed at the time when all target subjects underwent pre-treatment and interim F-18 FDG PET/CT scans.
  - Analyze correlation between imaging parameters and non-imaging biomarker such as NLR using Pearson or Spearman correlation analysis/ biserial correlation analysis
Correlation between biomarkers and treatment response | The primary analysis can be performed when all study subjects have elapsed more than 6 months after the start of treatment.
  - Analyze correlation between biomarkers and treatment response using Point-biserial correlation analysis
Correlation between biomarkers and patient prognosis | The primary analysis can be performed when all study subjects have elapsed more than 12 months after the start of treatment.
  - Analyze the correlation between biomarkers and prognosis (OS, PFS) using Cox proportional hazard model

CONTACTS AND LOCATIONS:
Overall Officials: hoyun lee, M.D., Ph.D., Principal Investigator — Samsung Medical Center, Department radiology
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Takada K, Toyokawa G, Yoneshima Y, Tanaka K, Okamoto I, Shimokawa M, Wakasu S, Haro A, Osoegawa A, Tagawa T, Oda Y, Nakanishi Y, Mori M. 18F-FDG uptake in PET/CT is a potential predictive biomarker of response to anti-PD-1 antibody therapy in non-small cell lung cancer. Sci Rep. 2019 Sep 16;9(1):13362. doi: 10.1038/s41598-019-50079-2. PMID 31527660
- [Background] Goldfarb L, Duchemann B, Chouahnia K, Zelek L, Soussan M. Monitoring anti-PD-1-based immunotherapy in non-small cell lung cancer with FDG PET: introduction of iPERCIST. EJNMMI Res. 2019 Jan 29;9(1):8. doi: 10.1186/s13550-019-0473-1. PMID 30694399
- [Background] Humbert O, Cadour N, Paquet M, Schiappa R, Poudenx M, Chardin D, Borchiellini D, Benisvy D, Ouvrier MJ, Zwarthoed C, Schiazza A, Ilie M, Ghalloussi H, Koulibaly PM, Darcourt J, Otto J. 18FDG PET/CT in the early assessment of non-small cell lung cancer response to immunotherapy: frequency and clinical significance of atypical evolutive patterns. Eur J Nucl Med Mol Imaging. 2020 May;47(5):1158-1167. doi: 10.1007/s00259-019-04573-4. Epub 2019 Nov 23. PMID 31760467
- [Background] Seban RD, Mezquita L, Berenbaum A, Dercle L, Botticella A, Le Pechoux C, Caramella C, Deutsch E, Grimaldi S, Adam J, Ammari S, Planchard D, Leboulleux S, Besse B. Baseline metabolic tumor burden on FDG PET/CT scans predicts outcome in advanced NSCLC patients treated with immune checkpoint inhibitors. Eur J Nucl Med Mol Imaging. 2020 May;47(5):1147-1157. doi: 10.1007/s00259-019-04615-x. Epub 2019 Nov 21. PMID 31754795